CLINICAL TRIAL: NCT03296865
Title: Effects of Kinesio Taping in Rectus Femoris Activity and Sit-to-stand Movement in Children With Unilateral Cerebral Palsy: Placebo-controlled, Repeated-measure Design
Brief Title: Taping in Children With Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adriana Neves Dos Santos (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor-Investigator, Adriana Neves Dos Santos, Professor, Reseacher, Universidade Federal de Santa Catarina
Organization: Universidade Federal de Santa Catarina (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: fapesc2012/10558-6
Record Dates: First submitted 2017-09-25; First posted 2017-09-28 (Actual); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Cerebral Palsy
Keywords: taping; functionality; rehabilitation; muscle activity; electromyography
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Intervention Model Description: We used a blinded and repeated-measure design, with the application of a placebo condition
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Children and the person that performed the evaluation were blind only to KT and placebo conditions, since they did not know if KT was tensioned were not. The person that performed data analysis was blind to all conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Without taping (No Intervention): Evaluations without taping
- Kinesio taping (Experimental): Kinesio taping was apllied only one time. It was removed after intervention.
  Interventions: Device: Kinesio taping
- Placebo (Placebo Comparator): Placebo was apllied only one time. It was removed after intervention.
  Interventions: Device: Kinesio taping

INTERVENTIONS:
Device: Kinesio taping — We applied a hypoallergenic, porous and adhesive tape of cotton (Kinesio Tex Gold) placed over Rectus Femoris muscle of the affected limb. Children were taped in accordance to Kenzo Kase's Kinesio manual. We used a facilitation technique, from muscle origin to insertion, in a Y shape. For KT condition: base of the KT strip 3cm below the anterior iliac spine, over the RF muscle until the upper edge of the patella and stretchered with 100% tension. For placebo condition: same technique without tension in the entire tape.
  We verified the immediate effect of KT/placebo. After the evaluation, KT/placebo was removed.
  Other Names: taping
  Arms: Kinesio taping; Placebo

SUMMARY:
Kinesio taping (KT) has been commonly used in rehabilitation in children with Unilateral Cerebral Palsy (UCP). However, there is a lack of studies that verified the effects of KT in CP. We aimed to verify the effects of KT in the performance of sit to stand movement (STS) in children with spastic UCP (USCP). A blinded, placebo and repeated-measure design was applied. The setting was the rehabilitation clinic of the university and care facilities. Eleven children, aged from 6 to 12 years old (10.5±-2.8 years), diagnosed with USCP, Gross Motor Function Classification System levels I and II were evaluated. KT was applied over rectus femoris (RF) muscle of the affected limb. We considered three taping conditions: KT, without KT (with tension) and placebo (KT without tension). Mean root mean square (mRMS) of RF; initial, final and peak angles, and range of motion of trunk, pelvis, hip, knee and ankles joints; and total duration of STS were considered. STS was evaluated from three seat heights, neutral (100%), lowered (80%) and elevated (120%). Mixed ANOVA test was applied for angular variables of hip, knee and ankle, and mRMS of RF. Repeated ANOVA was applied for angular variables of trunk and pelvis, total duration.

DETAILED DESCRIPTION:
We evaluated a non-probability convenience sample. Participants were recruited in the rehabilitation clinic of the university and care facilities, between July of 2013 and July of 2014.

Body structures and functions and functionality component of the International Classification of Functioning, Disability and Healthy, were evaluated. Muscle activity (electromyography) and trunk and lower limbs alignment (kinematics) were evaluated as body structures and functions measures. Time used to perform STS was used as functionality measure.

We evaluated sit to stand in three conditions: a) without taping; b) with KT, which was characterized as the use of KT with tension; c) placebo.

Baseline measurement: STS without taping. The child was seated in a seat with adjustable height, without shoes. Both feet were symmetrically positioned shoulder width apart and arms were crossed over the chest. The participants could not use their arms to push up off the chair. Also, the child should be seated with gluteal and the upper thighs regions supported in seat. Children performed STS in a speed that simulated the one usually adopted in daily routine.

Baseline measurement was evaluated in three seat heights: neutral, elevated and lowered. Neutral corresponded to a seated position with 90° of hip, knee and ankle flexion. Lowered and elevated were defined as, respectively, 80 and 120% of neutral height.The order of seat heights was randomized by drawing lots. A interval of 5 minutes was allowed between each seat height.

Evaluations were carried out in two testing episodes, with one-week interval between them. On the first day, additional to baseline, the child performed STS with KT or placebo. The determination of which tape condition would be applied was randomized by drawing lots. A 15-minute interval between baseline and tape condition was established. On the second day, the tape condition that was not performed on the first day was evaluated. In all conditions, the child performed STS in three seat heights.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with unilateral spastic Cerebral Palsy
* Aged from 6 and 12 years
* Ability to perform sit to stand movement without support in three seat heights

Exclusion Criteria:

* Ability to understand simple commands
* Muscle shortening in hamstrings, gastrocnemius and hip flexors
* Deformity in the lower limbs, such as fixed hip and knee flexion, that could compromise STS
* Surgical procedures in lower limbs and trunk in previous 12 months
* Botulinum toxin injection in lower limbs in the previous 6 months
* Not attending physical therapy at least 2 times a week during the last 6 months

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 11 (Actual)
Dates: Start 2014-03-01 (Actual); Primary Completion 2015-03-03 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Rectus femoris muscle activity | change measures (2 days, 3 measures)
  A portable surface electromyography (Trigno™ Wireless EMG System, DelSys®, Boston, USA) was used to evaluate RF activity (sampling 2400Hz).
  Electrode was positioned at RF of both limbs while the child was lying in supine. Skin preparation and electrode placement were performed according to SENIAM guidelines.
Trunk and lower limbs alignment (kinematics) | change measures (2 days, 3 measures)
  A six-camera motion analysis system Qualisys ProReflex MCU (QUALISYS-MEDICAL AB®, Gothenburg, Sweden) recorded body kinematics (sampling 240Hz). 27 non co-linear passive markers (15mm) were placed.
  Angular variation of trunk, pelvis, hip, knee and ankle were assessed using the Visual 3D software. We considered initial, final and peak angles. We also evaluated range of motion defined as the difference between final and initial angles.
Time used to perform sit to stand movement | change measures (2 days, 3 measures)
  Time in seconds from kinematics evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Nelci Adriana Cicuto Ferreira Rocha, Phd, Study Director — Universidade de São Carlos
Locations (1):
- Universidade Federal de São Carlos, São Carlos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary outcomes will be made available
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: One year after study completion